CLINICAL TRIAL: NCT05261646
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Two-Stage Phase Ⅲ Study Evaluating the Efficacy and Safety of Hetrombopag Olamine Tablets in Treatment of Chemotherapy-Induced Thrombocytopenia
Brief Title: A Clinical Study of Hetrombopag Olamine Tablets in Adults Receiving 21-day Cycles of Chemotherapy for Solid Tumours, Who Are Delayed for at Least 1 Week From Their Scheduled Cycle Because of Chemotherapy-induced Thrombocytopenia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-TPO-CIT-301
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-02

CONDITIONS: Chemotherapy-Induced Thrombocytopenia
MeSH Terms: interventions — hetrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hetrombopag (Experimental)
  Interventions: Drug: Hetrombopag
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Hetrombopag — Stage 1： Hetrombopag lower dose； Hetrombopag higher dose
  Stage 2:
  Hetrombopag X mg (dose to be determined based on Stage 1 results)
  Arms: Hetrombopag
Drug: Matching placebo — Matching placebo（Stage 1；Stage 2）
  Arms: Matching placebo

SUMMARY:
The study is aimed to evaluate the efficacy of different doses of hetrombopag compared to placebo, measured by the proportion of subjects that can complete two planned consecutive chemotherapy cycles with no modification of chemotherapy regimen (i.e., delayed start, dose reduction, omission, or discontinuation) because of thrombocytopenia [platelet count <100×109/L], to determine an optimal dose of hetrombopag and to demonstrate its superiority over placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female gender, age ≥18 years.
2. Histologically or cytologically confirmed solid tumor (e.g., non-small-cell lung carcinoma [NSCLC], breast, bladder, pancreatic, gastrointestinal, or colon/colorectal cancer).
3. Receiving a chemotherapy cycle of 21 days with one or more of the following chemotherapeutic drugs:

   * Antimetabolites, including gemcitabine, etc.
   * Platinum-based agents, including carboplatin, nedaplatin, cisplatin, and lobaplatin, etc.
   * Anthracyclines, including doxorubicin, daunorubicin, epirubicin, etc.
   * Alkylating agents, including cyclophosphamide, ifosfamide, etc.
4. Delay for at least 1 week from the scheduled chemotherapy cycle because of thrombocytopenia (PC <75×109/L for 4 weeks after the start of the previous chemotherapy cycle.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
6. Expected survival ≥ 6 months at screening.
7. At least 2 remaining chemotherapy cycles with current chemotherapy regimen.
8. Agreement for subjects of childbearing potential to take effective contraceptive measures throughout the study (including male or female condoms, contraceptive foam, contraceptive gel, contraceptive diaphragm, contraceptive cream, contraceptive suppository, abstinence, and inserted intrauterine devices, etc.); except female subjects who have undergone hysterectomy, bilateral salpingectomy, bilateral tubal ligation or have been in menopause for more than 1 year, and male subjects who have undergone bilateral vasectomy or ligation.
9. Signed ICF for voluntary participation in the study and good compliance.

Exclusion Criteria:

1. PC <25×109/L or ≥75 x 109/L at screening or enrollment.
2. Hematopoietic diseases other than CIT (e.g., primary immune thrombocytopenia).
3. Hematologic malignancies.
4. Thrombocytopenia caused by reasons other than chemotherapy, including but not limited to chronic liver disease, hypersplenism, infection, and hemorrhage, within 6 months before screening.
5. Intracranial metastases or disease.
6. Bone marrow involvement or bone marrow metastasis on routine imaging.
7. Conditions that require emergent treatment (e.g., superior vena cava syndrome, spinal cord compression).
8. Pelvic, spinal radiotherapy, or large-field bone radiation received within 3 months prior to screening.
9. Severe cardiovascular disorders or interventions within 6 months before screening: New York Heart Association (NYHA) Class III-IV; arrhythmias known to increase the risk of thromboembolism (e.g., atrial fibrillation); prolonged QTc (>450 msec for males and >460 msec for females); coronary artery angioplasty, stenting, or bypass grafting.
10. Any arterial or venous thrombosis (e.g., deep vein thrombosis, pulmonary embolism, transient ischemic attack/stroke, or myocardial infarction) within 6 months prior to screening.
11. Known bleeding disorders, platelet dysfunction.
12. Use of anticoagulants or non-steroidal anti-inflammatory drugs (NSAIDs) within 7 days of screening. The use of low dose aspirin (81 mg) is allowed.
13. Severe hemorrhage (e.g., gastrointestinal, or intracranial hemorrhage) within 2 weeks before screening.
14. Absolute neutrophil count (ANC) <1.5× 109/L, or Hb <80 g/L. Use of granulocyte colony stimulating factor, red blood cell, or erythropoietin infusion therapy that meets routine clinical practice is allowed.
15. Significantly abnormal liver function:

    * For subjects without liver metastasis: alanine aminotransferase/aspartate aminotransferase (ALT/AST) > 3 × ULN (upper limit of normal), TBL > 3 × ULN.
    * For subjects with liver metastases: ALT/AST ≥ 5 × ULN, TBL > 3 × ULN.
16. Abnormal renal function: estimated glomerular filtration rate (eGFR) ≤ 60 mL/min (Cockcroft-Gault estimated creatinine clearance).
17. Previous treatments with TPO-R agonists (e.g., eltrombopag, romiplostim) at any time before screening or enrollment.
18. Platelet transfusion received within 72 hours prior to screening or enrollment, with PC >75×109/L at screening or enrollment.
19. Known or expected allergy or intolerance to the active substances or excipients of hetrombopag.
20. Acute or chronic hepatitis C or hepatitis B.
21. Human immunodeficiency virus (HIV) infection.
22. Confirmed SARS-CoV-2 (COVID-19) infection (validated test positive), or suspected COVID-19 infection (clinical symptoms without documented test results) within 4 weeks before screening, or close contact with a person with known or suspected COVID-19 infection within 2 weeks before screening (subject may be included with a documented negative result for a validated COVID-19 test).
23. Pregnancy/intention to become pregnant during the study period or lactation.
24. Participation in another clinical trial within 30 days or 5 half-lives of an investigational product (whichever is longer) prior to screening.
25. Investigator's judgement that participation in the study creates a significant risk for the health of a subject, or his/her condition may affect evaluation of the safety and/or efficacy of hetrombopag.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of treatment "responders" who do not require modification of chemotherapy regimen because of thrombocytopenia (PC <100×109/L) during two planned consecutive chemotherapy cycles without the use of rescue treatment. | 56 days after the first dose of study drug
  Cochran-Mantel-Haenszel (CMH) test will be used to make a comparison between each hetrombopag group and the placebo group.

SECONDARY OUTCOMES:
Time to first platelet response, defined by PC ≥100×109/L. | 56 days after the first dose of study drug
  Will be analyzed by a log-rank test stratified by the randomization stratification factors.
  The Kaplan-Meier (KM) method will be used to describe the time-to-event data.
Proportion of subjects achieving PC ≥100×109/L. | 14 days after the first dose of study drug
  Will be analyzed with the CMH test
Time duration of PC ≥100×109/L. | 42 days after the start of the first chemotherapy cycle
  Will be analyzed with the log rank test and KM plots
PC nadir from the start of the first on-study chemotherapy cycle through the end of the double-blind treatment period. | 42 days after the start of the first chemotherapy cycle]
  An Analysis of Covariance (ANCOVA) will be used.
Time duration of severe thrombocytopenia, defined as a PC of 50×109/L | 56 days after the first dose of study drug
  Will be analyzed with the log rank test and KM plots.
Proportion of subjects without serious bleeding events, defined as grade ≥ 2, according to the World Health Organization Bleeding scale. | 56 days after the first dose of study drug
  Will be analyzed with the CMH test.
Proportion of subjects with at least single incidence of platelet transfusion or other rescue treatment. | 56 days after the first dose of study drug
  Will be analyzed with the CMH test.
Proportion of patients without chemotherapy regimen modifications due to any cause. | 14 days after the first dose of study drug
  Will be analyzed with the CMH test.
Number adverse events (AEs) as assessed by CTCAE v5.0. | up to 140 days of treatment with study drug plus 6 months of follow-up.
  Arithmetic summary statistics will be provided.

IPD SHARING:
Plan to Share IPD: Undecided